CLINICAL TRIAL: NCT04032132
Title: The Local Application of Curcumin in Conjunction With the Surgical Treatment of Intrabony Periodontal Defects "Controlled Clinical Study With Evaluation of Curcumin Release Profile"
Brief Title: Curcumin Paste as an Adjunctive Therapy in Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Gamal, Administrator of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FER16 20-M
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis
Keywords: curcumin; CBCT; HPLC; periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Curettage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- curcumin paste in conjunction with open flap debridement surge (Experimental): curcumin paste (2% circumin) in conjunction with open flap debridement surgery
  Interventions: Drug: curcumin paste; Procedure: curettage
- open flap debridement surgery only (Placebo Comparator): surgical treatment for periodontal pocket
  Interventions: Procedure: curettage

INTERVENTIONS:
Drug: curcumin paste — curcumin is a herb used for medical purpose
  Arms: curcumin paste in conjunction with open flap debridement surge
Procedure: curettage — open flab debridement surgery

SUMMARY:
The turmeric (Curcuma longa) plant, a herb belonging to the ginger family. The most active component of turmeric is curcumin, which makes up 2 to 5% of the spice. Curcumin showed has antibacterial effect against periodontal pathogen and positive result regarding conventional treatment of periodontal disease due to its anti-inflammatory, anti-oxidant and wound healing properties. This study will be carried out to examine the effect of curcumin when used in conjunction with open flap debridement treating deep periodontal pockets. (suggesting that it may have positive effect)

DETAILED DESCRIPTION:
The present study entailed twenty four patients having stage II or stage III, Grade A periodontitis with 24 intrabony defects. Patients were divided into two groups; group I was subjected to open flap debridement only. Group II was subjected to curcumin paste (2%curcumin)in conjunction with open flap debridement Clinical parameters including plaque index, sulcus bleeding index, probing depth and clinical attachment level were recorded pre-surgical. Moreover, radiographic examination was performed by cone beam computed tomography (CBCT) just before the surgery . Vertical bone defects were exposed by full thickness mucoperiosteal flap following intrasulcular incision and thorough debridement was performed. Group II received local application of curcumin paste.The same initial clinical parameters were recorded three and six months postoperatively. Radiographic measurements were recorded six months post surgically.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age range 25-45 years.
2. At least a single posterior 2-3 wall periodontal defect of pocket depth ≥ 5mm; clinical attachment level ≥ 3 mm, Intrabony component ≥ 3 mm and with plaque index ≤1 (Löe 1967) and bleeding index ≤1 (Mühlemann & Son 1971). All the previous criteria were determined 2 weeks after phase I conventional periodontal therapy.
3. Systemically Healthy as evidenced by Burket's oral medicine health history questionnaire (Glick et al., 2008).

Exclusion Criteria:

* 1- Smokers. 2- Pregnant. 3- Patient unwilling to comply to periodontaloral hygienic instructions. 4- Vulnerable groups. (e.g: Decisionally impaired individual)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-20 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
clinical score | change from base line at 6 months
  Evaluate the influence of curcumin paste on the clinical outcomes of the surgical treatment.to see if curcumin has a positive effect in reduction oh deep periodontal pockets and leads to greater bone gain

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, professor, Study Director — Faculty of dentistry -Ain Shams university

IPD SHARING:
Plan to Share IPD: No